CLINICAL TRIAL: NCT06104384
Title: Socio-demographics of Injury Insurance Claims by Chronic Pain Patients
Brief Title: Characteristics of Injury Claims by Chronic Pain Patients
Status: Recruiting | Type: Observational
Sponsor: Salem Anaesthesia Pain Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: SalemAne2018 Injury Claim Race
Record Dates: First submitted 2023-10-23; First posted 2023-10-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Social Functioning; Chronic Pain; Injuries; Disabilities Multiple
Keywords: Injury Claim; Disability Claim
MeSH Terms: conditions — Social Adjustment; Chronic Pain; Wounds and Injuries | interventions — Palliative Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult chronic pain patients: Adult chronic pain patients who received pain management
  Interventions: Behavioral: Behavioral and supportive therapy

INTERVENTIONS:
Behavioral: Behavioral and supportive therapy — Behavioral and supportive therapy

SUMMARY:
Chronic pain is associated with injuries and disabilities. This prospective observational study explores the injury or disability claims made by chronic pain patients. It evaluates the socio-demographics of the patient population. It explores the impact of pain clinic services on the patients' injury rehabilitation, insurance claim outcome, and socioeconomic situation.

DETAILED DESCRIPTION:
Chronic pain is associated with injuries, disabilities, psychological disorders, and unemployment. Chronic pain patients usually make insurance claims for injury, disability, and unemployment.

This prospective observational study explores the injury, disability, and compensation claims made by chronic pain patients. The study evaluates the socio-demographics of the patient population; including their gender, age, ethnicity, occupation, employment status, income, education level, family status, and home location. It explores the impact of pain clinic services on the patients' injury rehabilitation course, insurance claim outcome, and socioeconomic situation.

ELIGIBILITY:
Inclusion Criteria:

* adult chronic pain patients
* patients with injury claim

Exclusion Criteria:

* pediatric patients
* patients without injury claim

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult chronic pain patients who are undergoing treatment in a specialist pain clinic
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2018-01-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients who had injury insurance claims approved | 12 months
  Percentage of patients with successful insurance claim approval

CONTACTS AND LOCATIONS:
Overall Officials: Olumuyiwa Bamgbade, MD,FRCPC, Principal Investigator — Salem Anaesthesia Pain Clinic
Locations (1):
- Salem Anaesthesia Pain Clinic, Surrey, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No